CLINICAL TRIAL: NCT02213627
Title: Randomized, Multicentric and Prospective Clinical Trial to Check the Cost-effectiveness of Corifollitropin Alfa vs. Recombinant FSH and/or HP-hMG
Brief Title: Use of Corifolitropin Alfa in Oocyte Donors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IVI Madrid (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Responsible Party: Principal Investigator, Antonio Requena, MD, PhD, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403-MAD-013-AR
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Female Reproductive Problem; Infertility
Keywords: Corifollitropin alfa, recombinant FSH, HP-hMG, apoptosis, oocyte donation
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Corifollitropin alfa (Experimental): From day 2-3 of mense, a single 100 microgram dose of corifollitropin alfa is administered. Daily doses of 0.25 mg GnRH antagonist will start on day 6 of stimulation and a single dose of 0.2 mg of GnRH agonist will be administered for triggering final oocyte maturation.
  Interventions: Drug: Corifollitropin alfa
- Recombinant FSH (Experimental): From day 2-3 of mense, daily injections of 150 IU of recombinant FSH will be administered. Daily doses of 0.25 mg GnRH antagonist will start on day 6 of stimulation and a single dose of 0.2 mg of GnRH agonist will be administered for triggering final oocyte maturation.
  Interventions: Drug: Recombinant FSH
- HP-hMG (Experimental): From day 2-3 of mense, daily doses of 225 IU of HP-hMG will be administered. Daily doses of 0.25 mg GnRH antagonist will start on day 6 of stimulation and a single dose of 0.2 mg of GnRH agonist will be administered for triggering final oocyte maturation.
  Interventions: Drug: HP-hMG

INTERVENTIONS:
Drug: Corifollitropin alfa
  Other Names: Elonva 100 micrograms
  Arms: Corifollitropin alfa
Drug: Recombinant FSH
  Other Names: Puregon 50 IU
  Arms: Recombinant FSH
Drug: HP-hMG
  Other Names: Menopur 600 IU
  Arms: HP-hMG

SUMMARY:
The purpose of this study is to determine if corifollitropin alfa (long-term gonadotropin administration) is effective in a controlled ovarian stimulation protocol in oocyte donors compared to daily gonadotropin administration (recombinant FSH or HP-hMG)

DETAILED DESCRIPTION:
In recent years, increasingly advances have been developed in terms of controlled ovarian stimulation protocols. These improvements have also moved into the way of administration of the different treatments, and at present, with subcutaneous devices, it is possible to offer advantages such as the ability to ensure administration of the correct dose or modify the dose before charging.

Simplification of ovarian stimulation protocols can help to reduce physical stress of the donors and the cancellation rate. The need for daily injection does not worsen the degree of compliance, but it generates some anxiety related to the administration of the right dose and / or the possibility of making a unconsciously mistake . Innovations in delivery devices could help reduce the stress associated with the stimulation itself and improve the welfare of the donor. Given these considerations, the need to develop a stimulation protocol that reduces the physical and emotional burden of reproduction treatment is established.

Corifollitropin alfa molecule is a full-length recombinant FSH generating a sustained effect of stimulation; a single subcutaneous injection of this drug is able to replace the first seven injections of any daily FSH preparation, so finally, the result would be an overall decrease in the number of injections needed for the whole cycle. Pharmacological and pharmacodynamic characteristics of corifollitropin alfa could facilitate the design of simple stimulation protocols and the need for fewer resources when monitoring the donor, including fewer clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 years who meet the entry criteria for the IVI Donor Program:
* Weight < 60 Kg
* Women with at least 6 antral follicles per ovary
* Women who will fit the protocoo during the period of the study
* Women who give written consent to participate in the test

Exclusion Criteria:

* Women with basal antral follicle count above 20 or below 6.
* Women with comorbidities, in the judgement of the investigator, that may interfere with the trearment of ovarian stimulation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes and mature oocytes | 3 months

SECONDARY OUTCOMES:
Fertilization and implantation rates | 3 months
Drop-out rate and cancellation rate | 3 months
Cost-effectiveness analysis | 6 months
Endocrine profile in serum and follicular fluid | 3 months
Apoptosis rate in cumulus cells | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Requena, MD, PhD, Principal Investigator — IVI Madrid; Manuel Muñoz, MD, PhD, Study Chair — Instituto Valenciano de Infertilidad, IVI Alicante; Pilar Alamá, MD, PhD, Study Chair — IVI Valencia; María Cruz, PhD, Study Chair — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Madrid, Spain